CLINICAL TRIAL: NCT02103621
Title: Discontinuation of Long-term SRIs in Obsessive Compulsive Disorder
Brief Title: Assisting Obsessive Compulsive Disorder (OCD) Patients With Discontinuing Long-term Serotonin Reuptake Inhibitors (SRIs)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1402-002; 1R21MH100444-01A1 (NIH); 1402-002 (Other: Butler Hospital)
Record Dates: First submitted 2014-04-01; First posted 2014-04-04 (Estimated); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Obsessive Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Unifed Protocol (UP) for Discontinuation (Experimental): Unified Protocol (UP) for Discontinuation is delivered in 14 weekly individual sessions of 45-60 minutes followed by 3 booster sessions scheduled at two, four and eight weeks thereafter. The UP is a cognitive behavioral treatment that focuses on increasing emotional awareness and cognitive flexibility, preventing behavioral and emotional avoidance, and situational and interoceptive emotion-focused exposure. Participants will also receive 7 biweekly medication management sessions over 14 weeks with a study psychiatrist to facilitate gradual taper of SRI medication.
  Interventions: Behavioral: Unified Protocol (UP)
- Taper and Monitoring (TAP-M) (Active Comparator): Taper and Monitoring (TAP-M) is delivered in biweekly individual sessions over 14 weeks, with booster sessions at two, four, and eight weeks thereafter. TAP-M consists of assessment and monitoring. Participants will also receive 7 biweekly medication management sessions over 14 weeks with a study psychiatrist to facilitate gradual taper of SRI medication.
  Interventions: Behavioral: Taper and Monitoring (TAP-M)

INTERVENTIONS:
Behavioral: Unified Protocol (UP)
  Arms: Unifed Protocol (UP) for Discontinuation
Behavioral: Taper and Monitoring (TAP-M)
  Arms: Taper and Monitoring (TAP-M)

SUMMARY:
This study will address questions of fundamental clinical significance including: (1) whether OCD patients maintained on long term SRIs can be discontinued without symptom exacerbation, (2) whether trans-diagnostic cognitive-behavioral treatment will reduce worsening following discontinuation compared to Taper and Monitoring, and (3) whether predictors of successful SRI discontinuation can be identified.

ELIGIBILITY:
Inclusion Criteria:

1. 18 or older
2. Presence of mild to moderate OCD symptoms
3. Patient's treating clinician agrees that SRI discontinuation is clinically appropriate
4. Adequate trial of SRI (≥10 weeks) in the current treatment episode
5. Maintenance on SRI dose that has not increased due to significant clinical worsening in the two years prior to enrollment
6. English speaking

Exclusion Criteria:

1. Clinically significant suicidality or a suicide attempt within the past year
2. Presence of any clinical features warranting a higher level of care (partial or inpatient hospitalization)
3. Current or recent (past 6 months) alcohol or drug dependence or abuse
4. Current or past psychotic disorder or bipolar disorder
5. Moderate to severe depression, as indicated by a Hamilton Rating Scale for Depression (HRSD) (17-item) ≥ 14 or recent major depressive episode (past 6 months)
6. History of severe OCD (YBOCS ≥ 28)
7. Prior adverse experience with SRI discontinuation
8. Primary compulsive hoarding
9. Cognitive impairment that would interfere with study participation
10. Concomitant psychosocial treatment w/ proven efficacy in the treatment of OCD
11. Previous adequate trial of exposure-based treatment (e.g., history of 12 or more sessions) in past 5 years
12. Use of non-SRI psychotropic medications for OCD in the 3 months prior to enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-05; Primary Completion 2017-09 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Yale-Brown Obsessive Compulsive Scale (Y-BOCS) | 14 weeks post baseline

CONTACTS AND LOCATIONS:
Overall Officials: Christina L Boisseau, Ph.D., Principal Investigator — Butler Hospital
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States